CLINICAL TRIAL: NCT05319626
Title: Immediate Effects of Two Different Lower Limb Sensory Stimulation Strategies on Balance and Mobility in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sevim Beyza Ölmez, Principal Investigator, Gazi University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-844
Record Dates: First submitted 2022-03-28; First posted 2022-04-08 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Elderly; Balance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group 1 (Experimental): Compression socks with Textured insoles
  Interventions: Other: compression socks; Other: textured insoles
- Intervention group 2 (Experimental): Compression socks with Smooth insoles
  Interventions: Other: compression socks; Other: smooth insoles
- Intervention group 3 (Experimental): Smooth socks with Textured insoles
  Interventions: Other: textured insoles; Other: smooth socks
- Control group (Placebo Comparator): Smooth socks with Smooth insoles
  Interventions: Other: smooth socks; Other: smooth insoles

INTERVENTIONS:
Other: compression socks — The compression socks have a clinical pressure of 23-30 mm Hg. The socks are dressed to the participants based on the manufacturer's sizing guidelines.
  Arms: Intervention group 1; Intervention group 2
Other: textured insoles — The textured insoles have small, pyramidal peaks with centre-to-centre distances of approximately 2.5 mm (Evalite Pyramid EVA, 3 mm thickness, shore value A50, black). The insoles cut to a range of men's and women's standard EU shoe sizes. During the testing process, they are worn within a standardised shoe.
  Arms: Intervention group 1; Intervention group 3
Other: smooth socks — The smooth socks are a commercial stocking that does not have a compression feature, but has a similar thickness and color to the compression stocking. They have standard size.
  Other Names: control socks
  Arms: Control group; Intervention group 3
Other: smooth insoles — The smooth insoles have a completely flat surface (Evalite Pyramid EVA, 3 mm thickness, shore value A50, black). The insoles cut to a range of men's and women's standard EU shoe sizes. During the testing process, they are worn within a standardised shoe.
  Other Names: control insoles
  Arms: Control group; Intervention group 2

SUMMARY:
Falls are a major public health problem worldwide. As a result of changes in sensory system capacity with aging, postural control decreases and the risk of falling increases. Various lower-limb sensory stimulation strategies are applied to compensate for these changes in sensory system capacity. It has been determined that these practices can have positive effects on postural control. Among these stimulation strategies, compression stockings and textured insoles are frequently preferred because of their cost-effectiveness and ease of application. For these purpose, this study aims to examine the immediate effects of wearing textured insoles and compression stockings on balance and mobility in older adults. Thus, we will sight to discern whether interventions of the textured insoles and compression materials improve sensory afferent feedback in the foot.

DETAILED DESCRIPTION:
Within-subject experimental design with all participants tests under each of four randomly organized conditions: (i) Compression socks with textured insoles, (ii) Compression socks with smooth insoles, (iii) Smooth socks with textured insoles, (iv) Smooth socks with smooth insoles. With each condition, the participants are given a 5-minute warm-up period to get used to the insoles and stocking conditions, and then the testing process consisting of balance, mobility and foot sensation assessments is started. All data are collected randomly in a single testing session by the same researcher blind to the conditions.Before all data collection, each participant has a practice of test process to ensure familiarity with the devices and the procedures. A rest period of 10 minutes are given between applications.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults over the 65 years old with ability to stand independently without using any assistive devices
* No history of falls in the last 12 months
* Mini Mental State Examination (MMSE) score > 24 (normal)
* Berg Balance Test score > 40

Exclusion Criteria:

* Self-reported neurological, vestibular or neuromuscular diseases
* Current history of peripheral neuropathy
* Presence of severe visual impairment (such as cataracts or glaucoma)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Foot sensation test | in an average of one and half hour
  Foot plantar sense will be assessed with Semmes-Weinstein monofilament test. The foot sensation test will be performed (barefoot) immediately after each condition to determine the effect of the condition. 4 times in total.
Balance test | in an average of one and half hour
  Balance will be assessed using the Biodex-BioSway™ Portable Balance System, in different visual situations and support surfaces during bilateral standing. It will be measured with each condition, 4 times in total.
Mobility test | in an average of one and half hour
  Mobility will be assessed by selecting Time Up and Go and Walk parameters in the BTS G-Walk wearable motion analysis system. Time Up and Go test determines functional mobility, and fall risk. Walk test evaluates quantitative analysis for the performance of walking. It will be measured with each condition, 4 times in total.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Beyza Ölmez, Principal Investigator — Gazi University; Selda Başar, Study Director — Gazi University; Tuğçe Çoban, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woo MT, Davids K, Liukkonen J, Orth D, Chow JY, Jaakkola T. Effects of different lower-limb sensory stimulation strategies on postural regulation-A systematic review and meta-analysis. PLoS One. 2017 Mar 29;12(3):e0174522. doi: 10.1371/journal.pone.0174522. eCollection 2017. PMID 28355265
- [Background] Kenny RPW, Atkinson G, Eaves DL, Martin D, Burn N, Dixon J. The effects of textured materials on static balance in healthy young and older adults: A systematic review with meta-analysis. Gait Posture. 2019 Jun;71:79-86. doi: 10.1016/j.gaitpost.2019.04.017. Epub 2019 Apr 17. PMID 31022658
- [Background] Woo MT, Davids K, Chow JY, Jaakkola T. Acute effects of wearing compression knee-length socks on ankle joint position sense in community-dwelling older adults. PLoS One. 2021 Feb 8;16(2):e0245979. doi: 10.1371/journal.pone.0245979. eCollection 2021. PMID 33556067